CLINICAL TRIAL: NCT03413150
Title: Modeling of Amiodarone Effect on Heart Rate Control in Critically Ill Patients With Atrial Tachyarrhythmias
Acronym: AMIRA
Status: Completed | Type: Observational
Sponsor: Groupe Hospitalier Pitie-Salpetriere (Other)
Responsible Party: Principal Investigator, Joe Elie Salem, MD, Groupe Hospitalier Pitie-Salpetriere
Other Study IDs: CIC1421-17-13
Record Dates: First submitted 2018-01-22; First posted 2018-01-29 (Actual); Last update posted 2019-09-26 (Actual); Status verified 2019-09

CONDITIONS: Atrial Fibrillation; Atrial Tachycardia
MeSH Terms: conditions — Atrial Fibrillation | interventions — Amiodarone

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (1):
- severely ill patients receiving amiodarone for ATs: cohort study was conducted from January 2007 to April 2012 in the 18-bed medical ICU of a tertiary teaching hospital.Data were extracted from the files of 80 consecutive critically ill patients who had received at least one dose of amiodarone to treat or prevent atrial tachycardia during their hospitalization in the ICU.
  Interventions: Drug: Amiodarone

INTERVENTIONS:
Drug: Amiodarone — Data were extracted from the files of 80 consecutive critically ill patients who had received at least one dose of amiodarone to treat or prevent AT during their hospitalization in the ICU.

SUMMARY:
Aims Amiodarone is the gold-standard medication to control heart rate in critically ill patients with atrial tachyarrhythmias (ATs); however, effective doses and covariates influencing its efficacy remain unknown. The investigators therefore performed pharmacodynamic modeling of heart rate reduction induced by amiodarone in these patients. Methods and Results This observational study included 80 consecutive severely ill patients receiving amiodarone to treat ATs. A total of 1348 time-heart rate observations with 361 amiodarone dose administrations were analyzed during a period of up to 6 days after hospital treatment initiation using a nonlinear mixed-effect model. Pretreatment with amiodarone before intensive care administration, paroxysmal versus persistent AT, catecholamine infusion, and fluid and magnesium loading were among the covariates assessed in the model. In case of paroxysmal AT in a patient not pretreated with amiodarone, a 300 mg intravenous loading dose combined with an 800 mg oral dose on the first day, followed by 800 mg/day orally for 4 days was effective in achieving a heart rate between 80 and 115 bpm within the first day, and to maintain it during the next 4 days. Corresponding doses were twice as high in patients with persistent AT. Use of intravenous magnesium (p\0.02) and fluid loading (p\0.02) was associated with an earlier and greater heart rate decrease, while use of dobutamine had an opposite influence (p\0.05). Conclusions In critically ill patients with AT, the dose of amiodarone required to control heart rate is influenced by the type of AT and by other easily measurable conditions which may allow better individualization of amiodarone dosing.

ELIGIBILITY:
Inclusion Criteria:

* critically ill patients who had received at least one dose of amiodarone to treat or prevent AT during their hospitalization in the ICU.

Exclusion Criteria:

* Patients with paced rhythm or incomplete charts were excluded

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Critically ill patients who had received at least one dose of amiodarone to treat or prevent AT during their hospitalization from January 2007 to April 2012 in the 18-bed medical ICU of a tertiary teaching hospital
Sampling Method: Non-Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2007-01 (Actual); Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
Heart Rate | HR at 1rst administration of cordarone and then 4 to 6 times a day after each dosing until day 6 or death or ICU discharge
  HR was retrieved from patients ICU charts

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Nicot F, Procopi N, Nguyen LS. Intravenous amiodarone-induced acute liver failure in cardiac surgery intensive care unit. Therapie. 2018 Sep;73(4):355-357. doi: 10.1016/j.therap.2017.12.007. Epub 2017 Dec 30. No abstract available. PMID 29395301
- [Result] Artucio H, Pereira M. Cardiac arrhythmias in critically ill patients: epidemiologic study. Crit Care Med. 1990 Dec;18(12):1383-8. doi: 10.1097/00003246-199012000-00015. PMID 2245612
- [Result] Packer DL, Bardy GH, Worley SJ, Smith MS, Cobb FR, Coleman RE, Gallagher JJ, German LD. Tachycardia-induced cardiomyopathy: a reversible form of left ventricular dysfunction. Am J Cardiol. 1986 Mar 1;57(8):563-70. doi: 10.1016/0002-9149(86)90836-2. PMID 3953440
- [Result] Nerheim P, Birger-Botkin S, Piracha L, Olshansky B. Heart failure and sudden death in patients with tachycardia-induced cardiomyopathy and recurrent tachycardia. Circulation. 2004 Jul 20;110(3):247-52. doi: 10.1161/01.CIR.0000135472.28234.CC. Epub 2004 Jun 28. PMID 15226218
- [Result] European Heart Rhythm Association; European Association for Cardio-Thoracic Surgery; Camm AJ, Kirchhof P, Lip GY, Schotten U, Savelieva I, Ernst S, Van Gelder IC, Al-Attar N, Hindricks G, Prendergast B, Heidbuchel H, Alfieri O, Angelini A, Atar D, Colonna P, De Caterina R, De Sutter J, Goette A, Gorenek B, Heldal M, Hohloser SH, Kolh P, Le Heuzey JY, Ponikowski P, Rutten FH. Guidelines for the management of atrial fibrillation: the Task Force for the Management of Atrial Fibrillation of the European Society of Cardiology (ESC). Eur Heart J. 2010 Oct;31(19):2369-429. doi: 10.1093/eurheartj/ehq278. Epub 2010 Aug 29. No abstract available. PMID 20802247
- [Result] January CT, Wann LS, Alpert JS, Calkins H, Cigarroa JE, Cleveland JC Jr, Conti JB, Ellinor PT, Ezekowitz MD, Field ME, Murray KT, Sacco RL, Stevenson WG, Tchou PJ, Tracy CM, Yancy CW; ACC/AHA Task Force Members. 2014 AHA/ACC/HRS guideline for the management of patients with atrial fibrillation: executive summary: a report of the American College of Cardiology/American Heart Association Task Force on practice guidelines and the Heart Rhythm Society. Circulation. 2014 Dec 2;130(23):2071-104. doi: 10.1161/CIR.0000000000000040. Epub 2014 Mar 28. No abstract available. PMID 24682348
- [Result] Kumar A. Intravenous amiodarone for therapy of atrial fibrillation and flutter in critically ill patients with severely depressed left ventricular function. South Med J. 1996 Aug;89(8):779-85. doi: 10.1097/00007611-199608000-00005. PMID 8701376
- [Result] Clemo HF, Wood MA, Gilligan DM, Ellenbogen KA. Intravenous amiodarone for acute heart rate control in the critically ill patient with atrial tachyarrhythmias. Am J Cardiol. 1998 Mar 1;81(5):594-8. doi: 10.1016/s0002-9149(97)00962-4. PMID 9514456
- [Result] Mayr A, Knotzer H, Mutz N, Hasibeder W. Atrial tachyarrhythmia after cardiac surgery. Intensive Care Med. 1999 Feb;25(2):242-3. doi: 10.1007/s001340050827. No abstract available. PMID 10193563
- [Result] Galve E, Rius T, Ballester R, Artaza MA, Arnau JM, Garcia-Dorado D, Soler-Soler J. Intravenous amiodarone in treatment of recent-onset atrial fibrillation: results of a randomized, controlled study. J Am Coll Cardiol. 1996 Apr;27(5):1079-82. doi: 10.1016/0735-1097(95)00595-1. PMID 8609324
- [Result] Delle Karth G, Geppert A, Neunteufl T, Priglinger U, Haumer M, Gschwandtner M, Siostrzonek P, Heinz G. Amiodarone versus diltiazem for rate control in critically ill patients with atrial tachyarrhythmias. Crit Care Med. 2001 Jun;29(6):1149-53. doi: 10.1097/00003246-200106000-00011. PMID 11395591
- [Result] Carlsson J, Miketic S, Windeler J, Cuneo A, Haun S, Micus S, Walter S, Tebbe U; STAF Investigators. Randomized trial of rate-control versus rhythm-control in persistent atrial fibrillation: the Strategies of Treatment of Atrial Fibrillation (STAF) study. J Am Coll Cardiol. 2003 May 21;41(10):1690-6. doi: 10.1016/s0735-1097(03)00332-2. PMID 12767648
- [Result] Van Gelder IC, Hagens VE, Bosker HA, Kingma JH, Kamp O, Kingma T, Said SA, Darmanata JI, Timmermans AJ, Tijssen JG, Crijns HJ; Rate Control versus Electrical Cardioversion for Persistent Atrial Fibrillation Study Group. A comparison of rate control and rhythm control in patients with recurrent persistent atrial fibrillation. N Engl J Med. 2002 Dec 5;347(23):1834-40. doi: 10.1056/NEJMoa021375. PMID 12466507
- [Result] Donaldson L, Grant IS, Naysmith MR, Thomas JS. Acute amiodarone-induced lung toxicity. Intensive Care Med. 1998 Jun;24(6):626-30. doi: 10.1007/s001340050627. PMID 9681788
- [Result] Ratz Bravo AE, Drewe J, Schlienger RG, Krahenbuhl S, Pargger H, Ummenhofer W. Hepatotoxicity during rapid intravenous loading with amiodarone: Description of three cases and review of the literature. Crit Care Med. 2005 Jan;33(1):128-34; discussion 245-6. doi: 10.1097/01.ccm.0000151048.72393.44. PMID 15644659
- [Result] Papiris SA, Triantafillidou C, Kolilekas L, Markoulaki D, Manali ED. Amiodarone: review of pulmonary effects and toxicity. Drug Saf. 2010 Jul 1;33(7):539-58. doi: 10.2165/11532320-000000000-00000. PMID 20553056
- [Result] Lafont E, Urien S, Salem JE, Heming N, Faisy C. Modeling for critically ill patients: An introduction for beginners. J Crit Care. 2015 Dec;30(6):1287-94. doi: 10.1016/j.jcrc.2015.09.002. Epub 2015 Sep 4. PMID 26719063
- [Result] Tonet JL, Lechat P, Frank R, Lascault G, Fontaine G, Facquet J, Cohen A, Grosgogeat Y. [Electrocardiographic effects and antiarrhythmic action of 1200 mg of oral amiodarone per day]. Ann Cardiol Angeiol (Paris). 1984 Jul-Sep;33(5):309-15. French. PMID 6476769
- [Result] Kochiadakis GE, Igoumenidis NE, Solomou MC, Kaleboubas MD, Chlouverakis GI, Vardas PE. Efficacy of amiodarone for the termination of persistent atrial fibrillation. Am J Cardiol. 1999 Jan 1;83(1):58-61. doi: 10.1016/s0002-9149(98)00783-8. PMID 10073786
- [Result] Anastasiou-Nana M, Levis GM, Moulopoulos S. Pharmacokinetics of amiodarone after intravenous and oral administration. Int J Clin Pharmacol Ther Toxicol. 1982 Nov;20(11):524-9. PMID 7174155
- [Result] Pourbaix S, Berger Y, Desager JP, Pacco M, Harvengt C. Absolute bioavailability of amiodarone in normal subjects. Clin Pharmacol Ther. 1985 Feb;37(2):118-23. doi: 10.1038/clpt.1985.22. PMID 3967454
- [Result] Vardas PE, Kochiadakis GE, Igoumenidis NE, Tsatsakis AM, Simantirakis EN, Chlouverakis GI. Amiodarone as a first-choice drug for restoring sinus rhythm in patients with atrial fibrillation: a randomized, controlled study. Chest. 2000 Jun;117(6):1538-45. doi: 10.1378/chest.117.6.1538. PMID 10858380
- [Result] Lotto A, Satolli R, Baldini MR. Hemodynamic effects of amiodarone. Circulation. 1980 Sep;62(3):666. doi: 10.1161/01.cir.62.3.666. No abstract available. PMID 7398031
- [Result] Schwartz A, Shen E, Morady F, Gillespie K, Scheinman M, Chatterjee K. Hemodynamic effects of intravenous amiodarone in patients with depressed left ventricular function and recurrent ventricular tachycardia. Am Heart J. 1983 Oct;106(4 Pt 2):848-56. doi: 10.1016/0002-8703(83)90007-8. PMID 6613831
- [Result] Remme WJ, Kruyssen HA, Look MP, van Hoogenhuyze DC, Krauss XH. Hemodynamic effects and tolerability of intravenous amiodarone in patients with impaired left ventricular function. Am Heart J. 1991 Jul;122(1 Pt 1):96-103. doi: 10.1016/0002-8703(91)90764-9. PMID 2063768
- [Result] Jacqmin P, Snoeck E, van Schaick EA, Gieschke R, Pillai P, Steimer JL, Girard P. Modelling response time profiles in the absence of drug concentrations: definition and performance evaluation of the K-PD model. J Pharmacokinet Pharmacodyn. 2007 Feb;34(1):57-85. doi: 10.1007/s10928-006-9035-z. Epub 2006 Oct 19. PMID 17051439
- [Result] Evans SJ, Myers M, Zaher C, Simonson J, Nalos P, Vaughn C, Oseran D, Gang E, Peter T, Mandel W. High dose oral amiodarone loading: electrophysiologic effects and clinical tolerance. J Am Coll Cardiol. 1992 Jan;19(1):169-73. doi: 10.1016/0735-1097(92)90069-y. PMID 1729329
- [Result] Hainsworth R. Reflexes from the heart. Physiol Rev. 1991 Jul;71(3):617-58. doi: 10.1152/physrev.1991.71.3.617. No abstract available. PMID 2057525
- [Result] Fellahi JL, Parienti JJ, Hanouz JL, Plaud B, Riou B, Ouattara A. Perioperative use of dobutamine in cardiac surgery and adverse cardiac outcome: propensity-adjusted analyses. Anesthesiology. 2008 Jun;108(6):979-87. doi: 10.1097/ALN.0b013e318173026f. PMID 18497597
- [Result] Butterworth J. Dobutamine: too dangerous for "routine" administration? Anesthesiology. 2008 Jun;108(6):973-4. doi: 10.1097/ALN.0b013e318172fb98. No abstract available. PMID 18497594
- [Result] Miller S, Crystal E, Garfinkle M, Lau C, Lashevsky I, Connolly SJ. Effects of magnesium on atrial fibrillation after cardiac surgery: a meta-analysis. Heart. 2005 May;91(5):618-23. doi: 10.1136/hrt.2004.033811. PMID 15831645
- [Result] Mayr A, Ritsch N, Knotzer H, Dunser M, Schobersberger W, Ulmer H, Mutz N, Hasibeder W. Effectiveness of direct-current cardioversion for treatment of supraventricular tachyarrhythmias, in particular atrial fibrillation, in surgical intensive care patients. Crit Care Med. 2003 Feb;31(2):401-5. doi: 10.1097/01.CCM.0000048627.39686.79. PMID 12576943
- [Result] Kanji S, Williamson DR, Yaghchi BM, Albert M, McIntyre L; Canadian Critical Care Trials Group. Epidemiology and management of atrial fibrillation in medical and noncardiac surgical adult intensive care unit patients. J Crit Care. 2012 Jun;27(3):326.e1-8. doi: 10.1016/j.jcrc.2011.10.011. Epub 2012 Jan 4. PMID 22226423
- [Result] Singh BN, Singh SN, Reda DJ, Tang XC, Lopez B, Harris CL, Fletcher RD, Sharma SC, Atwood JE, Jacobson AK, Lewis HD Jr, Raisch DW, Ezekowitz MD; Sotalol Amiodarone Atrial Fibrillation Efficacy Trial (SAFE-T) Investigators. Amiodarone versus sotalol for atrial fibrillation. N Engl J Med. 2005 May 5;352(18):1861-72. doi: 10.1056/NEJMoa041705. PMID 15872201
- [Result] Sticherling C, Behrens S, Kamke W, Stahn A, Zabel M. Comparison of acute and long-term effects of single-dose amiodarone and verapamil for the treatment of immediate recurrences of atrial fibrillation after transthoracic cardioversion. Europace. 2005 Nov;7(6):546-53. doi: 10.1016/j.eupc.2005.05.017. Epub 2005 Sep 30. PMID 16216756
- [Result] Harris L, Hind CR, McKenna WJ, Savage C, Krikler SJ, Storey GC, Holt DW. Renal elimination of amiodarone and its desethyl metabolite. Postgrad Med J. 1983 Jul;59(693):440-2. doi: 10.1136/pgmj.59.693.440. PMID 6622326
- [Result] Vietti-Ramus G, Veglio F, Marchisio U, Burzio P, Latini R. Efficacy and safety of short intravenous amiodarone in supraventricular tachyarrhythmias. Int J Cardiol. 1992 Apr;35(1):77-85. doi: 10.1016/0167-5273(92)90058-b. PMID 1563883
- [Result] Brodsky MA, Allen BJ, Walker CJ 3rd, Casey TP, Luckett CR, Henry WL. Amiodarone for maintenance of sinus rhythm after conversion of atrial fibrillation in the setting of a dilated left atrium. Am J Cardiol. 1987 Sep 1;60(7):572-5. doi: 10.1016/0002-9149(87)90307-9. PMID 3630939
- [Result] Kochiadakis GE, Igoumenidis NE, Parthenakis FI, Chlouverakis GI, Vardas PE. Amiodarone versus propafenone for conversion of chronic atrial fibrillation: results of a randomized, controlled study. J Am Coll Cardiol. 1999 Mar 15;33(4):966-71. doi: 10.1016/s0735-1097(98)00678-0. PMID 10091823
- [Result] Greenberg ML, Lerman BB, Shipe JR, Kaiser DL, DiMarco JP. Relation between amiodarone and desethylamiodarone plasma concentrations and electrophysiologic effects, efficacy and toxicity. J Am Coll Cardiol. 1987 May;9(5):1148-55. doi: 10.1016/s0735-1097(87)80320-0. PMID 3571754
- [Result] Deharo JC, Durand A, Macaluso G, Malaterre H, Le Tallec L, Panagides D, Bory M, Djiane P. Clinical electrophysiologic effects of a single high oral dose of amiodarone. Fundam Clin Pharmacol. 1997;11(3):275-80. doi: 10.1111/j.1472-8206.1997.tb00196.x. PMID 9243260
- [Result] Patsilinakos S, Christou A, Kafkas N, Nikolaou N, Antonatos D, Katsanos S, Spanodimos S, Babalis D. Effect of high doses of magnesium on converting ibutilide to a safe and more effective agent. Am J Cardiol. 2010 Sep 1;106(5):673-6. doi: 10.1016/j.amjcard.2010.04.020. Epub 2010 Jul 23. PMID 20723644
- [Result] Salem JE, Dureau P, Funck-Brentano C, Hulot JS, El-Aissaoui M, Aissaoui N, Urien S, Faisy C. Effectiveness of heart rate control on hemodynamics in critically ill patients with atrial tachyarrhythmias managed by amiodarone. Pharmacol Res. 2017 Aug;122:118-126. doi: 10.1016/j.phrs.2017.06.004. Epub 2017 Jun 10. PMID 28610957
- [Result] Salem JE, El-Aissaoui M, Alazard M, Hulot JS, Aissaoui N, Le-Heuzey JY, Funck-Brentano C, Faisy C, Urien S. Modeling of Amiodarone Effect on Heart Rate Control in Critically Ill Patients with Atrial Tachyarrhythmias. Clin Pharmacokinet. 2016 Aug;55(8):991-1002. doi: 10.1007/s40262-016-0372-9. PMID 26946135